CLINICAL TRIAL: NCT05025891
Title: Reducing Inequalities in Access to Care in French Guiana: ISe-santé, a Randomized Study Evaluating a Model for Implementing E-health in the Management of HIV
Brief Title: ISe-santé, a Study Evaluating a Model for Implementing E-health in the Management of HIV Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ISe-SANTE
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: HIV; Telemedicine
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: control (No Intervention): Patients continue consultations as usual in HDJA or at UMIT.
- Arm 2: teleconsultation alone (Experimental): Patients are directed to the tele-monitoring platform without specific accompaniment.
  Interventions: Other: Teleconsultation
- Arm 3: teleconsultation and mediation (Experimental): Patients are referred to the tele-monitoring platform with specific support with mediation.
  Interventions: Other: Teleconsultation

INTERVENTIONS:
Other: Teleconsultation — Patients are randomized into groups in which there are either teleconsultations alone or with the help of a mediator to carry out their follow-up care
  Arms: Arm 2: teleconsultation alone; Arm 3: teleconsultation and mediation

SUMMARY:
It is a randomized, controlled, open-label, parallel group study of 3 arms, among patients followed for chronic HIV infection at Cayenne hospital. The main objective of the study is to evaluate the effectiveness of follow-up of these patients by teleconsultation associated or not with health mediation.

DETAILED DESCRIPTION:
The COVID-19 pandemic crisis has strained health systems, and chronic disease monitoring has often been put on hold, without yet really measuring the resulting health impact. In this context, e-Health has benefited from considerable momentum to overcome the shortcomings that have arisen, to allow remote monitoring of patients infected with COVID 19, to protect patients and caregivers and avoid nosocomial infections. Telemedicine is all the more relevant in Guyana as there are issues of geographic isolation, lack of specialists and critical mass of health professionals. In French Guiana, faced with the arrival of teleconsultation tools, a fear of professionals is their applicability for the most vulnerable populations, not knowing how to read or speak French and having restricted access to digital technology. Moreover HIV infection is an ever stigmatizing infection affecting populations that are often extremely precarious, requiring specialist monitoring and lifelong treatment.

The study team propose to carry out a randomized, controlled, open-label, parallel group study of 3 arms, among patients followed for chronic HIV infection at Cayenne hospital : 1/ Control group with classic follow-up at Cayenne hospital. 2/Teleconsultation only group: patients referred to the remote monitoring platform without specific support. 3/Teleconsulation group + mediator: patients referred to the remote monitoring platform with support from a health mediator Patients will be followed every 3 months or 6 months depending on the judgment of the investigating physician for 12 months in the study (primary endpoint evaluated at 1 year). Number of patients to be included: 450 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HIV infection.
* Patient with a regular follow-up for more than three months in the adult day hospital or in the infectious diseases department of the Cayenne Hospital Center.
* Patient of legal age.
* Patient having signed the consent form..

Exclusion Criteria:

* Pregnant patient
* Patient with a severe neurological or psychiatric history (significant cognitive disorders, intellectual disability).
* Patient with a physical disability that prevents communication via the e-Health platform (mute patient, visually and hearing impaired, specific manual motor disability, bedridden patient).
* Patient who does not master one of the languages available at the mediation.
* Patients under guardianship or trusteeship, people under protective measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-09-04 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportions of patients who followed the schedule proposed by the physician at inclusion (or revised during important events) in the 3 arms. | The inclusion period (1 year)

SECONDARY OUTCOMES:
Identification of the best strategy for implementing an e-Health platform in French Guiana in the management of chronic HIV infection | The inclusion period (1 year)
The proportion of patients throughout the inclusion period (1 year) likely to use the platform will be assessed using the number of patients meeting the inclusion criteria (having agreed to participate in the research or not). | The inclusion period (1 year)
The obstacles to the use of an e-health platform will be evaluated using a questionnaire for caregivers and patients and based on the number of failed connections | The inclusion period (1 year)
Patient satisfaction score assessed with study specific questionnaire | The inclusion period (1 year)
Caregiver satisfaction score assessed with study specific questionnaire | The inclusion period (1 year)
Evaluation of the material needs to guarantee accessibility of the consultation places | The inclusion period (1 year)
Evaluation of the material needs for the implementation and maintenance of the e-health platform | The inclusion period (1 year)
Measurement of the average intervention time of the doctors per patient | The inclusion period (1 year)
Measurement of the average intervention time of the mediators per patient | The inclusion period (1 year)
Measurement of the average intervention time of the ETP nurse per patient | The inclusion period (1 year)
Compare the patients followed up with the platform and the patients followed up in classic consultation on: the proportion of check-ups done during the same duration of follow-up, the proportion of patients with an undetectable viral load, the proportion | The inclusion period (1 year)
proportion of check-ups done during the same duration of follow-up between patients followed up with the platform and the patients followed up in classic consultation | The inclusion period (1 year)
proportion of patients with an undetectable viral load between patients followed up with the platform and the patients followed up in classic consultation | The inclusion period (1 year)
Questionnaire for all the care providers assessed with study specific questionnaire | The inclusion period (1 year)
  In order to evaluate the number of patients lost to follow-up, service congestion, patient waiting time, knowledge of the patient's pathway, communication with the patient, the number of missed consultations and the viral load of patients followed via the platform.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided